CLINICAL TRIAL: NCT03787238
Title: GM-18 - A Randomized, Multicenter, Study for the prEvention and Acute Treatment of Migraine Using Open Label Non-invasive Vagal Nerve Stimulation, Versus Standard of Care (REAL)
Brief Title: A Randomized, Multicenter, Study for the prEvention and Acute Treatment of Migraine (REAL)
Acronym: REAL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Company decision
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GM-18
Record Dates: First submitted 2018-12-20; First posted 2018-12-26 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- non-invasive Vagus Nerve Stimulation (Experimental): nVNS (non-invasive vagus nerve stimulation) treatment with the gammaCore Sapphire device and standard of care
  Interventions: Device: non-invasive vagus nerve stimulation
- Standard of Care (No Intervention): Standard of Care treatment

INTERVENTIONS:
Device: non-invasive vagus nerve stimulation — non-invasive vagus nerve stimulation using the gammaCore Sapphire device
  Arms: non-invasive Vagus Nerve Stimulation

SUMMARY:
This is a randomized study for the prevention and acute treatment of migraine using open label nVNS and standard of care versus standard of care.

.

DETAILED DESCRIPTION:
A randomized study for the prevention and acute treatment of migraine using open label nVNS and standard of care versus standard of care.

Eligible subjects will participate in a 4 week run-in period after which they will be randomized (1:1) to either nVNS and standard of care (nVNS group) or standard of care (SOC group) for 12 weeks. The nVNS group will use the nVNS device preventatively and acutely for the treatment of migraine. The SOC group will continue to use their regular standard of care migraine treatment medications for the duration of the 12 week randomized period.

ELIGIBILITY:
Inclusion Criteria:

* Is 18 years of age or above.
* Has been previously diagnosed with episodic or chronic migraine (with or without aura) in accordance with the ICHD-3 Classification criteria.
* Experience at least 6 and no more than 24 headache days per month and a minimum of 4 migraine attacks per month (over the last 3 months).
* Has age of onset of migraine less than 50 years old.
* Stable regime for any migraine preventative medications for the last 3 months and agrees to maintain stable regime for duration of the study.
* Agrees to and in clinician opinion is able to use the nVNS device as intended, follow all of the requirements of the study including follow-up visit requirements, record required study data in the subject dairy, and other self-assessment questionnaires.
* Availability of internet/Web access for Web-based e-diary completion
* Is able to provide written Informed Consent.

Exclusion Criteria:

* Requires use of oral or injectable steroids for concomitant medical condition that in the opinion of the investigator will interfere with the study.
* Has a history of any intracranial aneurysm, intracranial haemorrhage, brain tumour or significant head trauma.
* Has a structural abnormality at the nVNS treatment site (e.g. lymphadenopathy previous surgery or abnormal anatomy).
* Has pain at the nVNS treatment site (e.g. dysesthesia, neuralgia and/or cervicalgia).
* Has other significant pain problem (e.g. cancer pain or other head or facial disorder) that in the opinion of the investigator may confound the study assessments
* Has known or suspected severe cardiac disease (e.g. symptomatic coronay artery disease, prior myocardial infarction, congestive heart failure (CHF)).
* Has known or suspected severe cerebrovascular disease, (e.g. prior stroke or transient ischemic attack, symptomatic carotid artery disease, prior cartoid endarterectomy or other vascular neck surgery).
* Has known or suspected own and/or family history of cardiac disease (including but not limited to ischemic heart disease, rhythm disturbances, congenital abnormalities cardiac myopathies), or presents risk factors strongly associated with risk for developing cardiologic abnormalities that in the opinion of the investigator might compromise subjects safety using n-VNS.
* Has had a cervical vagotomy.
* Has uncontrolled high blood pressure (systolic >160 diastolic > 100 after 3 repeated measurements within 24 hours).
* Is currently implanted with an electrical and/or neurostimulator device (e.g. cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, cochlear implant, Spehnopalatine ganglion stimulator or Occiptial nerve stimulator).
* Has been implanted with metal cervical spine hardware or has a metallic implant near the nVNS stimulation site (e.g. in the head, neck of thorax).
* Presents a suspicion of secondary headache.
* Previous diagnosis of medication overuse headache within the last 3 months
* Has a history of syncope (within the last 1 year).
* Has a history of seizures (within the last 1 year).
* Has a known or suspicion of substance abuse or addiction (within the last 1 year).
* Has initiated medications for migraine prophylaxis in the previous 30 days, or in the case of Botulinum toxin and monoclonal antibodies against CGRP injections in the previous 90 days.
* Has failed an adequate trial (two months or greater) of at least 3 classes of a drug therapy for the prophylaxis of migraine.
* Is pregnant or of childbearing years and is unwilling to use and accepted form of birth control (condom or contraceptive pill).
* Is participating in any other therapeutic clinical investigation or has participated in a clinical trial in the preceding 30 days.
* Belongs to a vulnerable population or has any condition such that his or her ability to provide informed consent, comply with the follow-up requirements, or provide self- assessments is compromised (e.g. homeless, developmentally disabled and prisoner).
* Has previously used the gammaCore device within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-15 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in number of migraine days during the last four weeks in the twelve-week randomized period compared with the four-week run-in period | The last four weeks in the randomization period compared to the four week run-in period.
  Reduction in number of migraine days during the last four weeks in the twelve-week randomized period compared with the four-week run-in period

SECONDARY OUTCOMES:
Reduction in number of headache days during the last four-weeks in the twelve-week randomized period compared to the four-week run-in period | The last four weeks in the randomization period compared to the four week run-in period.
  Reduction in number of headache days during the last four-weeks in the twelve-week randomized period compared to the four-week run-in period
Reduction in number of migraine days and headache days (separately) | 12 week randomised period
  Reduction in number of migraine days and headache days (separately) during weeks 1 through 4, 5 through 8 in the 12 week randomised period
Rate of responders for the nVNS group compared to the standard of care group. | The last four weeks in the randomization period compared to the four week run-in period.
  Rate of responders (mean reduction in migraine days during the last four weeks in the twelve-week randomization period compared to the four-week run-in period dichotomized as <25% vs. ≥25%, <50% vs ≥50% and <75% vs ≥75%, separately) for the nVNS group compared to the standard of care group.
Acute treatment response for nVNS and standard of care therapies | 12 week randomised period
  Acute treatment response for nVNS and standard of care therapies at 30, 60 and 120 minutes post-treatment, for all treated migraine attacks in the twelve-week randomized period
Consistency of response | 12 week randomised period
  Consistency of response as defined as the percentage of subjects who achieve treatment response in 25%, 50% and 75% or greater of their attacks, in subjects treating at least two attacks, for nVNS and standard of care therapies for all treated migraine attacks during the randomized period
Safety and tolerability of nVNS as measured by adverse events | 12 week randomised period
  Safety and tolerability of nVNS as measured by adverse events

OTHER OUTCOMES:
Change in acute headache medication use | 12 week randomization period compared to the four week run-in period
  Change in acute headache medication use (proportion of attacks with acute medication use prior to or at 120 minutes post-treatment) for all treated attacks in the twelve-week randomized period compared to the four week run-in period in the nVNS group
Presence or absence of nausea, vomiting, photophobia, phonophobia | 12 week randomised period
  Presence or absence of nausea, vomiting, photophobia, phonophobia at 0, 30, 60 and 120 minutes post treatment for nVNS and standard of care therapies for all treated migraine attacks in the randomized period

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Sinclair, MD, Principal Investigator — University of Birmingham
Locations (17):
- Danish Headache Center, Glostrup Municipality, Denmark
- Germany (4):
  - CTC, University Medical Center Hamburg-Eppendorf, Hamburg
  - Migräne- und Kopfschmerzklinik Königstein, Königstein im Taunus
  - Klinik für Neurologie, Ludwig-Maximilliams-Universität, Klinikum Grosshadern, München
  - Klinik und Poliklinik für Neurologie, Universitätsmedizin Rostock, Rostock
- Italy (4):
  - National Neurological Institute C. Mondino Foundatio, Mondino, Pavia
  - U.O. Neurologia III - Cefalee e Neuroalgologia, Fondazione IRCCS Istituto, Milan
  - Department of Neurological, Motor and Sensorial Sciences, IRCCS San Raffaele, Rome
  - University of Turin, Turin
- Spain (4):
  - Headache Unit, University Hospital Vall d'Hebron, Barcelona
  - Servicio de Neurologia, Hospital Ruber Internacional, Madrid
  - Servicio de Neurologia, Clinica Universidad de Navarra, Pamplona
  - Servicio de Neurologia, Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (4):
  - Hull Royal Infirmary, Neurology Department, Hull, East Yorkshire
  - University of Birmingham, Birmingham
  - Queen Elizabeth Hospital Queen, Gateshead
  - Sunderland Royal Hospital, Sunderland